CLINICAL TRIAL: NCT02604875
Title: The Circadian Rhythm of Copeptin
Acronym: Co-Rhythm
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKNZ 2015-266
Record Dates: First submitted 2015-11-10; First posted 2015-11-16 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Circadian Rhythm; Copeptin Blood Levels
MeSH Terms: interventions — Observation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- observational: Blood samples will be taken for measuring copeptin levels in healthy subjects.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — blood sampling during 24 hours

SUMMARY:
The circadian rhythm of copeptin will be examined in healthy subjects.

DETAILED DESCRIPTION:
In 18 healthy volunteers the circadian rhythm of copeptin will be examined by withdrawing blood samples for copeptin levels every 30 minutes for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* acute illness
* chronic illness
* pregnancy
* Anemia defined as Hb < 30g/l

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
measurement of copeptin values in mmol/l within 24 hours to assess the amount of release in a day curve. | 24 hours
  The primary outcome measure is to compare the copeptin concentration in the early afternoon and the early morning by blood sampling at different time points. Evaluation of the question if there is a circadian rhythm in the copeptin release.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, MD, Prof., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No